CLINICAL TRIAL: NCT00073463
Title: A Multicenter, Double-Blind, Placebo Controlled, Phase II Study of Aerosolized tgAAVCF for the Treatment of Cystic Fibrosis
Brief Title: Safety and Efficacy of Recombinant Adeno-Associated Virus Containing the CFTR Gene in the Treatment of Cystic Fibrosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Targeted Genetics Corporation (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25E01; RAC-0301-569
Record Dates: First submitted 2003-11-21; First posted 2003-11-25 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Cystic Fibrosis
Keywords: Gene Transfer; Pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Genetic: tgAAVCF

SUMMARY:
The purpose of this study is to confirm the improvement in pulmonary function and cytokine levels observed in the recently completed multidose aerosol study for the treatment of Cystic Fibrosis (CF).

DETAILED DESCRIPTION:
Cystic Fibrosis is an autosomal recessive disorder with an incidence of approximately 1 in 33000 live births. It is due to defects in the CFTR gene, which is located on chromosome 7. Gene Therapy holds the promise of addressing the primary defect in CF by reconstituting the CFTR function in the lung. tgAAVCF, which has been genetically engineered to contain the CFTR gene, has been extremely well tolerated following single and multiple dose administrations to the nose, sinus, and lung. Dose-dependent gene transfer has been demonstrated. Although vector gene expression has not been detected, evidence consistent with biological activity was observed in maxillary sinus study, and statistically significant changes in the FEV1 and IL-8 levels were observed in the recently completed multidose aerosol study. These findings are worthy of further investigation.

ELIGIBILITY:
Eligible subjects will be randomized to two aerosolized doses of either tgAAVCF or placebo 30 days apart. Subjects will undergo pulmonary function testing every two weeks during the active portion of the study (three months) and will be followed for safety for a total of seven months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - UAB-Childrens Health System, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - UC San Diego, San Diego, California
  - University of Colorado-The Childrens Hospital, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Childrens Hospital, Boston, Massachusetts
  - The Minnesota CF Center, Minneapolis, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania